CLINICAL TRIAL: NCT04081493
Title: The Efficacy of Low-load Blood Flow Restricted Resistance Exercise in Patients With Knee Osteoarthritis Scheduled for Total Knee Arthroplasty: A Multicenter, Randomized Controlled Trial
Brief Title: The Efficacy of Low-load Blood Flow Restricted Resistance Before TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Okklusionsprojektet
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Total Knee Replacement
Keywords: Low-load blood flow restricted exercise; Preconditioning; Functional capacity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (BFRE) (Experimental): Low-load blood flow restricted exercise 3/weekly for 8 weeks before TKR 10-min warm-up followed by unilateral leg press and unilateral knee extension
  Interventions: Other: Low-load blood flow restricted exercise
- Group 2 (CON) (No Intervention): No training before TKR

INTERVENTIONS:
Other: Low-load blood flow restricted exercise — Leg press and knee extension exercise 3 times per week for 8 weeks. Repetition scheme: 30-15-15-until exhaustion interspaced by 30 sec rest. 5 min "free-flow" rest between exercises
  Arms: Group 1 (BFRE)

SUMMARY:
The primary aim of this study is to investigate the efficacy of 8 weeks of Low-load blood flow restricted exercise (BFRE) compared to receiving standard care only (no preoperative training) before total knee replacement (TKR) on postoperative 30-seconds chair stand test (30s-CST). We hypothesize that 8 weeks of preoperative BFRE will increase chair stand performance 3 months postoperatively. Secondary aims are to investigate the efficacy of 8 weeks of preoperative BFRE compared to receiving standard care only on changes in muscle strength 3 months after TKR and investigate associations to functional capacity and quality of life. Furthermore, it will be investigated if 8 weeks of BFRE induces muscle hypertrophy and increases satellite cell and myonuclei content of the vastus lateralis muscle.

DETAILED DESCRIPTION:
BFRE is resistance training with low loads (30% 1repetition maximum (RM) performed with concurrent partial blood flow restriction by means of pneumatic cuff compression around the working limb.

Group 1 (BFRE):

BFRE group: Will perform 3/weekly supervised BFRE sessions for 8 weeks from a physiotherapist educated in administering BFRE. Each session will consist of a 10-min warm up followed by two different unilateral lower-limb resistance training exercises: leg press and knee extension. Each exercise will be performed with the affected lower limb only and consist of 4 rounds interspaced by 30 seconds of rest. 1st round: 30 repetitions (reps); 2nd round: 15 reps; 3rd round: 15 reps; 4th round: until exhaustion. Between each exercise the patients will rest for 5 minutes without blood flow restriction.

Patients will rest in a standardized resting position between each set to maintain the desired resting cuff-pressure.

The occlusion pressure will be set at 60% of total limb occlusion pressure and starting load intensity will be 30% 1repetition maximum (1RM) in both exercises. If patients can perform more than 15 repetitions in the 4th exercise set, the exercise load will be increased with the minimum extra load possible.

Group 2 (control Group):

CON group: Will follow standard procedures before a TKA and be encouraged to live their lives as usual up until TKA.

The study is a multicenter (2 sites), randomized (allocation 1:1), assessor blinded, controlled trial Outcomes will be measured at baseline (9-10 weeks before surgery), in the week of surgery and 3- and 12 months postoperatively. Muscle biopsies will be taken from all patients undergoing surgery at Horsens Regional Hospital. Muscle biopsies will be taken at baseline, during surgery and 3 months postoperatively.

The 12 months follow-up assessment will be analyzed and presented in papers during a subsequent Post Doc-period.

All patients will be scheduled to receive TKR and receive a standard multimodal surgical program with standardized perioperative care. Specifically, all patients will be invited to a preoperative information meeting 2-3 weeks prior to surgery where nurses, surgeons, and physiotherapists will be providing detailed information about pain management, nutrition, the surgical procedure (i.e. basic knowledge about a prosthesis, risks related to smoking, restrictions related to living with a TKR, long-term results, and living with a TKR), physical activity, postoperative home-based rehabilitation, load-management, etc.

On the day of surgery patients will be hospitalized at one of the two orthopedic departments and TKR procedures will be performed by an orthopedic surgeon. The day after surgery patients will be trained once or twice per day by a physiotherapist towards fulfilling the following discharge criterions: independency in in-and-out of bed and sit-to-stand activities, independency in walking and stair-negotiation with crutches, ADL activities, and home-based exercises during the hospitalization period. Patients will generally be discharged within ~1-2 days after fulfilling all the above discharge criteria. After discharge, all patients will receive a standard home-based rehabilitation program aimed at increasing knee mobility and lower extremity muscle strength. However, if considered necessary by the physiotherapist in charge of the patient, patients can receive additional supervised knee-specific exercise therapy at private physiotherapy clinics, municipal rehabilitation centers, or specialized hospital-based rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 50 years scheduled for TKA at Horsens- or Silkeborg Regional Hospital.

Exclusion Criteria:

* Severe cardiovascular diseases (New York Heart Association class III and IIII), previous stroke incident, thrombosis incident
* Traumatic nerve injury in affected limb
* Unregulated hypertension (Systolic ≥180 or diastolic ≥110 mmHg)
* Spinal cord injury
* Pregnancy
* Planned other lower limb surgery within 12 months
* Cancer diagnosis and currently undergoing chemo-, immuno-, or radiotherapy
* Inadequacy in written and spoken Danish
* an existing prosthesis in the index limb
* living more than 45 minutes from either Horsens Regional Hospital or Silkeborg Regional Hospital.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
30-seconds chair stand test (30-sec CST) | change in 30-sec CST from baseline to 3 months after surgery
  The 30s-CST measures the number of sit-to-stand repetitions completed within 30 seconds. Patients will be instructed to perform a sit-to-stand movement starting from a seated position (seat height 43 cm without armrests) having the feet placed flat on the floor shoulder width apart, and arms crossed on chest to a standing position (hip and knee joints fully extended) repeated as many times as possible for 30 seconds.

SECONDARY OUTCOMES:
Timed Up & Go | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  The TUG assesses the time required for patients to stand from a chair (seat height 46 cm) walk around a tape mark 3 meters away and sit into the chair at return.
4x10 meter fast-paced walk test (40m-FWT) | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  The 40m fast-paced walk test (40m-FWT) measures the total time taken to walk 4 x 10 m excluding turns (meter/sec).
1RM leg press strength | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  1 Repetition maximum (RM) is the maximal load (kg) a patient is able to concentrically press in the leg press machine. The 1RM will be estimated from a 5-8RM leg press test. The 1RM will be calculated as [1RM = load (kg)/1.0278-0.0278·number of repetitions)
1RM knee extension strength | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  1 Repetition maximum (RM) is the maximal load (kg) a patient is able to concentrically lift in the knee extension machine. The 1RM will be estimated from a 5-8RM leg press test. The 1RM will be calculated as [1RM = load (kg)/1.0278-0.0278·number of repetitions)
Isometric knee extensor strength | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  Isometric knee extensor muscle strength will be assed with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table.
Isometric knee flexor strength | Measured at baseline, in the week of surgery, 3 months after surgery, and 12 months after surgery
  Isometric knee flexor muscle strength will be assed with the participants seated on a examination table with knees and hip positioned at 90 degree flexion. Assessment of muscle strength will be performed with a hand-held dynamometer, fixed with an adjustable rigid belt to the examination table.
Muscle biopsy sampling and analysis - myofiber morphology (cross sectional area, fiber type composition, myonuclei number) and myogenic stemm cell (satellite cell) content | Measured at baseline, in the week of surgery, and 3 months after surgery
  needle biopsies (100-150 mg) will be obtained from the vastus lateralis muscle of patients undergoing TKR at Horsens Regional Hospital
Knee disability and Osteoarthritis Outcome Score (KOOS) | Measured at baseline, in the week of surgery, 6 weeks after surgery, 3 months after surgery, and 12 months after surgery
  KOOS is a patient-administered knee specific questionnaire comprising five subscales Pain; Symptoms; Activities of daily living; Sport & Recreation; and Knee-Related Quality of Life.
EuroQol Group 5-dimension (EQ-5D-5L) | Measured at baseline, in the week of surgery, 6 weeks after surgery, 3 months after surgery, and 12 months after surgery
  The EQ-5D-L5 is a self-completion questionnaire consisting of two parts; first part of the EQ-5D-5L comprises five dimensions involving mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Adverse events | 3 months after surgery
  Adverse events will be defined as unpredicted or unintended events, signs, or disease occurring during the period from inclusion until the 3-month follow-up (primary end-point) resulting in contact with the healthcare system (hospital or general practitioner) independent of whether or not the event is related to the intervention or outcome assessments

OTHER OUTCOMES:
Blood pressure (used for eligibility) | Baseline
  Blood pressure will be measured with an electronic commercial blood pressure device
Exercise compliance and progression | The exercise period (8 weeks)
  project physiotherapists will register compliance with the BFRE sessions and progression during all 8 weeks for the patients in the BFRE Group.
Numeric Rating Scale Pain (NRS pain) | Baseline, during each training session, in the week of surgery, 3 months after surgery, 12 months after surgery
  The NRS for pain is a segmented unidimensional 11-item measure of pain intensity in adults
Declining to be operated | 3 months after surgery
  At 3 months follow up patients will be asked whether they decided to be operated or not
Postoperative supervised physiotherapy | 6 weeks after surgery, 3 months after surgery, 12 months after surgery
  Any participation in postoperative supervised training will be attained at all follow-up assessments by using patient-reported questionnaires (yes/no; type of exercise) in both the BFRE group and the CON group
Knee joint range of motion | baseline, in the week of surgery, 3 months after surgery, 12 months after surgery
  Patients knee joint range of motion will be measured using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Stian L Jørgensen, MSc, Principal Investigator — Department of Physio and Occupational Therapy, Horsens Regional Hospital; Inger Mechlenburg, DMSc, PhD, Study Director — Department of Clinical Medicine, Aarhus University, Denmark; Per Aagaard, Prof, PhD, Study Director — Department of Sports Science and Clinical Biomechanics; Marie B Bohn, PhD, Study Director — Department of Orthopaedic Surgery
Locations (3):
- Denmark (3):
  - Aarhus University Hosspital, Aarhus, Aarhus N
  - Horsens Regional Hospital, Horsens
  - Silkeborg Regional Hospital, Silkeborg

IPD SHARING:
Plan to Share IPD: Yes
Horsens Regional is responsible for handling all personal data provided by both sites in accordance to the Clinical Trial Agreement and the EU General Data Protection Regulation (GDPR)
Access Criteria: Silkeborg Regional Hospital and Aarhus University Horspital agree that information directly related to the protocol and trial, including data, material, Intellectual Property and results generated from the trial shall be the property of Horsens Regional Hospital, and shall be treated in strict confidence, and shall not be disclosed to any third party, or use for its benefit or the benefit of any third party, without the prior written consent of Horsens Regional Hospital, except for data that is (i) publicly known or available from other sources who are not under a confidentially obligation to the other party; (li) has been made available by the other party without confidentiality obligation; or (iii) is independently developed or otherwise already known by or available to the other party without a confidentiality obligation; or (iv) is already required disclosed by law.

REFERENCES:
- [Derived] Jorgensen SL, Aagaard P, Bohn MB, Hansen P, Hansen PM, Holm C, Mortensen L, Garval M, Tonning LU, Mechlenburg I. The Effect of Blood Flow Restriction Exercise Prior to Total Knee Arthroplasty on Postoperative Physical Function, Lower Limb Strength and Patient-Reported Outcomes: A Randomized Controlled Trial. Scand J Med Sci Sports. 2024 Nov;34(11):e14750. doi: 10.1111/sms.14750. PMID 39461901
- [Derived] Langgard Jorgensen S, Mechlenburg I, Bagger Bohn M, Aagaard P. Sit-to-stand power predicts functional performance and patient-reported outcomes in patients with advanced knee osteoarthritis. A cross-sectional study. Musculoskelet Sci Pract. 2024 Feb;69:102899. doi: 10.1016/j.msksp.2023.102899. Epub 2023 Dec 17. PMID 38141496
- [Derived] Jorgensen SL, Bohn MB, Aagaard P, Mechlenburg I. Efficacy of low-load blood flow restricted resistance EXercise in patients with Knee osteoarthritis scheduled for total knee replacement (EXKnee): protocol for a multicentre randomised controlled trial. BMJ Open. 2020 Oct 1;10(10):e034376. doi: 10.1136/bmjopen-2019-034376. PMID 33004382